CLINICAL TRIAL: NCT01804205
Title: Effects of Magnesium Sulphate on the Pharmacodynamics of Rocuronium in Patients 60 Years or Older: Randomised and Double-Blind Study
Brief Title: Magnesium Sulphate and Rocuronium in Patients Over 60
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pedro Rotava (Other Government)
Collaborators: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor-Investigator, Pedro Rotava, Mr, Instituto Nacional de Cancer, Brazil
Organization: Instituto Nacional de Cancer, Brazil (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MgRoc 60
Record Dates: First submitted 2013-02-28; First posted 2013-03-05 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Head and Neck Cancer
Keywords: magnesium sulfate; rocuronium; neuromuscular block; onset time; elderly
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulfate group (Experimental): In the magnesium group, patients received MgSO4 30 mg/kg in 0.9% physiological saline (total volume 100 ml) intravenously, for 10 min, and then continuous intravenous infusion of MgSO4 at a rate of 1 g/h during the surgical procedure until the maximum of 3 h.
  Interventions: Drug: Magnesium Sulfate
- Control group (Placebo Comparator): Controls received 100 ml of 0.9% physiological saline, for 10 min, and then continuous intravenous infusion of saline at a rate of 33 ml/h during the surgical procedure until the maximum of 3 h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — MgSO4 30 mg/kg in 0.9% physiological saline (total volume 100 ml) intravenously, for 10 min, and then continuous intravenous infusion of MgSO4 at a rate of 1 g/h during the surgical procedure until the maximum of 3 h
  Arms: Magnesium sulfate group
Drug: Placebo — 100 ml of 0.9% physiological saline, for 10 min, and then continuous intravenous infusion of saline at a rate of 33 ml/h during the surgical procedure until the maximum of 3 h
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the effects of MgSO4 administration on the pharmacodynamics of rocuronium in patients with 60 or more years of age.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* ASA physical status I-III
* Scheduled for elective oncologic head and neck surgery

Exclusion Criteria:

* Severe renal insufficiency (calculated creatinine clearance < 30 ml/min)
* Pre-operatory serum magnesium values > 2.5 mEq/l
* Patients receiving medications known to affect neuromuscular function (furosemide, aminoglycoside, anticonvulsivants, calcio channel blocker, litium, azatioprine, cyclofosfamide)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total recovery time of neuromuscular block (DurTOF0.9) | Within the surgical procedure
  Time from the start of injection of rocuronium until TOF ratio 0.9

SECONDARY OUTCOMES:
Onset time | Within the surgical procedure
  Time from the start of injection of rocuronium until 95% depression of the first twitch (T1) of the TOF
Clinical duration (Dur25%) | Within the surgical procedure
  Time from the start of injection of rocuronium until T1 of the TOF had recovered to 25% of the initial T1 value
Recovery index (Dur25-75%) | Within the surgical procedure
  Time between 25% and 75% recovery of the initial T1 value
Recovery time (Dur25%TOF0.9) | Within the surgical procedure
  Time between 25% recovery of the initial T1 value and a TOF ratio of 0.9

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Rotava, MD, Principal Investigator — Instituto Nacional de Cancer
Locations (1):
- Instituto Nacional de Câncer, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Kussman B, Shorten G, Uppington J, Comunale ME. Administration of magnesium sulphate before rocuronium: effects on speed of onset and duration of neuromuscular block. Br J Anaesth. 1997 Jul;79(1):122-4. doi: 10.1093/bja/79.1.122. PMID 9301400
- [Background] Czarnetzki C, Lysakowski C, Elia N, Tramer MR. Time course of rocuronium-induced neuromuscular block after pre-treatment with magnesium sulphate: a randomised study. Acta Anaesthesiol Scand. 2010 Mar;54(3):299-306. doi: 10.1111/j.1399-6576.2009.02160.x. Epub 2009 Nov 16. PMID 19919585
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Dubois PE, Gourdin M, Jamart J, Broka SM, Eucher P, D'Hollander A. Early and late parameters describing the offset of neuromuscular blockade are highly intercorrelated. Acta Anaesthesiol Scand. 2012 Jan;56(1):76-82. doi: 10.1111/j.1399-6576.2011.02596.x. PMID 22150409
- [Derived] Rotava P, Cavalcanti IL, Barrucand L, Vane LA, Vercosa N. Effects of magnesium sulphate on the pharmacodynamics of rocuronium in patients aged 60 years and older: A randomised trial. Eur J Anaesthesiol. 2013 Oct;30(10):599-604. doi: 10.1097/EJA.0b013e328361d342. PMID 23635996